CLINICAL TRIAL: NCT07325630
Title: IBI363 Combined Chemotherapy for Perioperative Treatment of MHC-II-Negative Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: A Single-Center, Single-Arm Phase II Clinical Study
Brief Title: Perioprative Study of IBI363 in Patients With MHC-II-Negative Locally Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Party Secretary of the Clinical Research Institute, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI363Y122
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: IBI363 + Chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): IBI363 combination with oxaliplatin and capecitabine (XELOX) or S-1 and oxaliplatin (SOX) for perioprative treatment of locally advanced gastric and gastroesophageal junction adenocarcinoma
  Interventions: Drug: IBI363 + chemotherapy

INTERVENTIONS:
Drug: IBI363 + chemotherapy — IBI363 Q3W +XELOX Q3W (Oxaliplatin 130 mg/m2, IV, Q3W, Capecitabine ,1000mg/ m2, PO, Bid, d1-14, Q3W) or IBI363 Q3W +SOX (Oxaliplatin 130 mg/m2, IV, Q3W, S-1, 40-60mg,PO, Bid, d1-14，Q3W )

SUMMARY:
This is a phase 2 study designed to evaluate the safety and efficacy of IBI363 in combination with oxaliplatin and capecitabine (XELOX) or S-1 and oxaliplatin (SOX) in perioprative treatment of locally advanced MHC-II-negative gastric and gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients voluntarily enrolled in this study and signed informed consent forms;
2. Age 18-75 years;
3. Pathologically confirmed gastric adenocarcinoma or gastroesophageal junction adenocarcinoma;
4. MHC-II negative, with <5% tumour cells displaying staining <2+ (grade 2 or stronger);
5. Clinically staged as cT3-4aN+M0 gastric or gastroesophageal junction adenocarcinoma confirmed by CT and/or laparoscopy (per AJCC 8th Edition staging);
6. No prior antineoplastic therapy for current disease (e.g., surgery, radiotherapy, chemotherapy, targeted therapy, immunotherapy);
7. Scheduled for surgical intervention following completion of neoadjuvant therapy;
8. Able to swallow tablets orally;
9. ECOG performance status 0-1;
10. Expected survival ≥6 months.

Key Exclusion Criteria:

1. Pregnant or lactating women, or women planning to become pregnant within 6 months prior to, during, or after the last dose of the investigational medicinal product.
2. Known signs of active bleeding from a lesion.
3. Patients with known dMMR/MSI-H status.
4. Oesophageal or pyloric near-obstruction affecting the subject's ability to eat or gastric emptying, or difficulty swallowing tablets.
5. Subjects with unresolved Grade >1 toxicity related to any prior antineoplastic therapy (excluding persistent Grade 2 alopecia, anaemia, peripheral neuropathy, electrolyte abnormalities correctable with treatment, or endocrine abnormalities controlled and stable with hormone replacement therapy).
6. Known dihydropyrimidine dehydrogenase (DPD) deficiency (or prior fluorouracil-containing therapy resulting in Grade 3 or higher mucositis).
7. Known hypersensitivity to any monoclonal antibody or component of the chemotherapy agents (capecitabine, oxaliplatin) (resulting in Grade 3 or higher hypersensitivity reaction).
8. History of epileptic seizures, active, newly diagnosed, or untreated central nervous system metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal metastases.
9. Clinically significant cardiovascular or cerebrovascular disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate of ITT population | Up to 3 years
  The proportion of subjects in the cohort defined as having no residual tumour cells detected microscopically and lymph node-negative following neoadjuvant therapy.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) Rate or surgical population | Up to 3 years
  The proportion of subjects undergoingvradical surgery who, following neoadjuvant therapy, were found to have no residual tumour cells under microscopic examination and negative lymph nodes.
Major Pathologic Response (MPR) Rate of ITT Population | Up to 3 years
  The proportion of subjects in the enrolled population who achieved pathological residual tumour ≤10% as defined by tumour regression induced by neoadjuvant therapy.
Major Pathologic Response (MPR) Rate of surgical population | Up to 3 years
  The proportion of subjects undergoing radical surgery who achieved pathological residual tumour ≤10% following neoadjuvant therapy-induced tumour regression.
R0 Resection Rate | Up to 3 years
  The proportion of subjects defined as having undergone R0 resection within the radical resection population.
Event-free Survival (EFS) | Up to 3 years
  Defined as the time from randomization to the first occurrence of disease progression determined using RECIST v1.1, inoperable disease, local recurrence following surgery, distant metastasis, or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 3 years
  Defined as the time from randomization to death from any cause.
AE | Up to 90 days post last dose
  Number of participants experiencing clinical adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided